CLINICAL TRIAL: NCT06699836
Title: A Phase Two Study Evaluating Two Doses of Leronlimab (Pro 140) In Combination With Trifluridine + Tipiracil (TAS-102) + Bevacizumab in Participants With CCR5+, Microsatellite Stable (MSS), Relapsed Refractory Metastatic Colorectal Cancer (mCRC)
Brief Title: A Phase 2 Study of Leronlimab in Combination With TAS-102 + Bevacizumab in Previously Treated Participants With mCRC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CytoDyn, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CD-O-101
Record Dates: First submitted 2024-11-19; First posted 2024-11-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: Microsatellite Stable; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — leronlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 350 mg dose of leronlimab in combination with Trifluridine + Tipiracil (TAS-102) + Bevacizumab (Experimental): 350 mg dose of leronlimab in combination with Trifluridine + Tipiracil (TAS-102) + Bevacizumab
  Interventions: Drug: 350 mg leronlimab
- 700 mg dose of leronlimab in combination with Trifluridine + Tipiracil (TAS-102) + Bevacizumab (Experimental): 700 mg dose of leronlimab in combination with Trifluridine + Tipiracil (TAS-102) + Bevacizumab
  Interventions: Drug: 700 mg leronlimab

INTERVENTIONS:
Drug: 350 mg leronlimab — Leronlimab (PRO) 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5)
  Other Names: PRO 140
  Arms: 350 mg dose of leronlimab in combination with Trifluridine + Tipiracil (TAS-102) + Bevacizumab
Drug: 700 mg leronlimab — Leronlimab (PRO) 140 is a humanized IgG4, monoclonal antibody (mAb) to the C-C chemokine receptor type 5 (CCR5)
  Other Names: PRO 140
  Arms: 700 mg dose of leronlimab in combination with Trifluridine + Tipiracil (TAS-102) + Bevacizumab

SUMMARY:
This is an open label, randomized, two arm, multi-center study to explore the effect of leronlimab on the overall response rate/ overall survival and safety and tolerability when used in combination with trifluridine and tipiracil + bevacizumab in patients with CCR5+, MSS, mCRC who have progressed on prior treatment before participating in the study. The main questions this study aims to answer are:

1. Can leronlimab, in combination with standard of care therapies trifluridine and tipiracil+ bevacizumab, increase the objective response rate in persons with CCR5+, MSS, mCRC who have progressed on prior treatment before participating in the study.
2. Is leronlimab safe and well tolerated in these subjects when used in combination with standard of care therapies trifluridine and tipiracil+ bevacizumab.

DETAILED DESCRIPTION:
This is an open label, randomized, two arm, multi-center study to explore the effect of leronlimab on the overall response rate/ overall survival and the safety and tolerability when used in combination with trifluridine and tipiracil + bevacizumab in patients with CCR5+, MSS, relapsed refractory, mCRC who have been previously treated with fluoropyrimidine, oxaliplatin, and irinotecan-based chemotherapy, an anti-VEGF therapy, and, if RAS wild-type and medically appropriate, an anti-EGFR therapy.

This study will enroll approximately 60 participants, 30 participants in each of two arms evaluating either 350 mg or 700 mg of leronlimab, who are 18 years of age or older, with histologically confirmed metastatic colorectal cancer that is microsatellite stable (MSS) and CCR5+ (confirmed by an immunohistochemistry (IHC) assay). Participants will be randomized 1:1 to each arm, where approximately 30 participants will receive 350 mg of leronlimab + trifluridine and tipiracil + bevacizumab and approximately 30 will receive 700 mg of leronlimab + trifluridine and tipiracil + bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects age ≥ 18 years with a history of treated colorectal cancer with unresectable metastases of the primary colorectal cancer to other organs.
2. If HIV-1 positive, viral load must be < 50 copies/ml and participant must be on stable ART for at least 3 months.
3. Demonstrate positive tumor expression of CCR5 by IHC.
4. Adult patients with metastatic colorectal cancer (mCRC) who have been previously treated with fluoropyrimidine-, oxaliplatin-, and irinotecan-based chemotherapy, an anti-VEGF therapy, and, if RAS wild-type and medically appropriate, an anti-EGFR therapy.
5. Histologically confirmed for microsatellite stable MSS colorectal cancer by PCR, Immunohistochemistry (IHC) or Next-generation sequencing (NGS).
6. Have measurable disease per RECIST 1.1
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Expected survival of at least three months
9. No anti-cancer treatment within the last four weeks or at least 5 half-lives prior to treatment (except for palliative radiation therapy from which the patient has recovered from all adverse events).
10. Patients must have adequate organ and bone marrow function within 28 days prior to registration, defined as:

    i. Acceptable liver function:
    1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN) OR direct bilirubin ≤ ULN for participants with total bilirubin levels > 1.5 × ULN
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for participants with liver metastases).

    ii. Acceptable renal function:

    a) GFR ≥ 30 mL/min iii. Acceptable hematologic status:
    1. Hemoglobin ≥ 9 g/dL Note: Criteria must be met without packed red blood cell (pRBC) transfusion within the prior 2 weeks. Participants can be on stable dose of erythropoietin (≥ approximately 3 months).
    2. White blood cells > 2500/µL
    3. Absolute neutrophil count > 1500/µL
    4. Platelet count > 100 000/µL.
11. Clinically normal resting 12-lead ECG at Screening Visit or, if abnormal, considered not clinically significant by the Principal Investigator.

    a) No QTC interval exceeding 460 milliseconds (ms) for females, no QTC interval exceeding 450 ms for males.
12. Both male and female patients and their partners of childbearing potential must agree to use two medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], or one of the following methods of birth control (intrauterine devices, tubal sterilization or vasectomy) or must practice complete abstinence from intercourse of reproductive potential from study entry to 6 months after the last day of treatment (excluding women who are not of childbearing potential and men who have been sterilized).
13. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening Visit and negative urine pregnancy test prior to receiving the first dose of study.
14. Male participants must agree to use contraception and refrain from donating sperm for at least 120 days after the last dose of study intervention.
15. Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study.

Exclusion Criteria:

1. Known severe hypersensitivity towards monoclonal antibodies.
2. Clinically significant active coronary heart disease and cardiovascular insufficiency with hypotension (systolic blood pressure <100 mmHg) per PI discretion
3. Prior history of other malignancies, except early-stage prostate cancer or basal cell carcinoma that has been surgically resected.
4. Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test) or hepatitis C or known viral infections.
5. Are pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the Screening Visit through 120 days after the last dose of study intervention.
6. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
7. Stroke and/or transient ischemic attack within 6 months prior to screening.
8. Placement of a cardiac stent or bypass surgery within 6 months of screening
9. Tumor invasion of a large vascular structure (e.g., pulmonary artery, superior or inferior vena cava).
10. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

    Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
11. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
12. Inability to follow protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of leronlimab in combination with trifluridine and tipiracil + bevacizumab in participants with CCR5+, refractory, MSS, mCRC. | From enrolment through end of treatment at 12 months
  Efficacy will be measured as the effect on objective response rate (ORR) of leronlimab when used in combination with trifluridine and tipiracil + bevacizumab in patients with CCR5+, refractory, MSS, mCRC.
  ORR is defined as the proportion of subjects with the best overall response (BOR) or confirmed CR or confirmed PR according to RECIST version 1.1.

SECONDARY OUTCOMES:
To assess the safety and tolerability of leronlimab when used in combination with trifluridine and tipiracil + bevacizumab in patients with CCR5+, refractory, MSS, mCRC. | From enrolment through end of treatment at 12 months.
  Treatment Emergent AE's (TEAE) are defined as events with an onset on or after the first treatment. TEAEs will be summarized by treatment group, System Organ Class, and preferred term. The following TEAE summaries will be provided:
  * All TEAEs
  * TEAEs related to study drug.
  * All TEAEs by severity
  * Serious TEAEs
  * Serious TEAEs related to study drug.
  * TEAE reported in 5% or more participants in any treatment group.
  * TEAEs leading to discontinuation of study treatment.
  * TEAEs leading to interruption of study treatment.
  * TEAEs leading to death.
To assess the duration of response of leronlimab in combination with trifluridine and tipiracil + bevacizumab in participants with CCR5+, MSS, mCRC | From enrolment through end of treatment at 12 months.
  The time from the first documentation of response, either partial or complete, to the documentation of the objective tumor progression or until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - City of Hope Orange County Lennar Foundation Cancer Center, Irvine, California
  - Pacific Hematology Oncology Associates, San Francisco, California
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Summit Cancer Center, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Undecided